CLINICAL TRIAL: NCT02112760
Title: Specific Stabilization Exercise With Ultrasound Feedback For Patient With Recurrent Low Back Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Collaborators: National Health Research Institutes, Taiwan (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 200903075R
Record Dates: First submitted 2014-04-10; First posted 2014-04-14 (Estimated); Last update posted 2014-04-14 (Estimated); Status verified 2014-04

CONDITIONS: Recurrent Low Back Pain
Keywords: specific stabilization exercise; ultrasound; low back pain
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Patient (Experimental): To evaluate the effect of specific stabilization intervention in recurrent low back pain participants
  Interventions: Other: specific stabilization exercise

INTERVENTIONS:
Other: specific stabilization exercise — The specific stabilization exercise refers to an exercise that targets the deep trunk muscle, including the multifidus and transversus abdominis with ultrasound feedback.

SUMMARY:
1. Specific aim 1:Identify factors that influence muscle performance by use of ultrasound imaging.

   Hypothesis: Gender, age, and BMI affect the muscle performance of deep trunk muscles.
2. Specific aim 2. To compare the performance of trunk deep muscles (transversus abdominis and multifidus) and the sensation and pain thresholds of patients with recurrent low back pain with asymptomatic subjects.

   Hypothesis: patients with recurrent low back pain have:

   (A) less activation of the transversus abdominis and multifidus, (B) peripheral and central sensitization, with decreased sensation and pain thresholds in the lumbar and foot areas.
3. Specific aim 3. To determine the performance of the transversus abdominis and multifidus, and the sensation and pain thresholds by use of ultrasound feedback training in asymptomatic adults, and to compare these results with the traditional training protocols for trunk stabilization.

   Hypothesis: Specific stabilization exercise using ultrasound feedback training is more effective in activating deep trunk muscles and increasing sensation and pain thresholds than the traditional stabilization training protocol in asymptomatic adults.
4. Specific aim 4. To determine the performance of the transversus abdominis and multifidus, and the sensation and pain thresholds by using the ultrasound feedback training in adults with low back pain, and to compare these results with the traditional training protocols for trunk stabilization.

Hypothesis: Specific stabilization exercise using ultrasound feedback training is more effective in activating deep trunk muscles and increasing sensation and pain thresholds than the traditional stabilization training protocol in adults with low back pain.

ELIGIBILITY:
Inclusion Criteria:

* recurrent low back pain for at least the past year
* lumbar region discomfort more than one day in the past three months
* recurrent discomfort more than one time in the past three months

Exclusion Criteria:

* pregnancy
* carcinoma
* systematic disease (rheumatic arthritis, ankylosing spondylitis etc)
* had surgery on lumbar region or lower extremities
* neurological symptom on lower extremities(numbness, pain etc)
* spondylolisthesis

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 72 (Actual)
Dates: Start 2011-06; Primary Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Increased change of sliding of transversus abdominis muscle and change of thickness on multifidus muscle in asymptomatic and low back pain group | pre treatment (0 week), post treatment(6 week)

SECONDARY OUTCOMES:
Decrease cold sensation threshold on left back and hot sensation threshold on left leg in both group | pre treatment (0 week), post treatment(6 week)

CONTACTS AND LOCATIONS:
Overall Officials: Shwu-Fen Wang, Ph.D, Study Director — chool of Physical Therapy, National Taiwan University
Locations (1):
- School of Physical Therapy, National Taiwan University, Taipei, ZhongZeng District, Taiwan